CLINICAL TRIAL: NCT00698243
Title: A Phase 1 Dose-escalation Study of Intermittent, Once Weekly, and Continuous Daily Oral OSI-027 Dosing in Patients With Advanced Solid Tumors or Lymphoma
Brief Title: Study of Oral OSI-027 in Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-027-101; 2007-006158-25 (EudraCT Number)
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Any Solid Tumor or Lymphoma
Keywords: OSI-027; Solid tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — OSI 027

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Schedule 1 (Experimental): Once daily for 3 days every 7 days
  Interventions: Drug: OSI-027
- Schedule 2 (Experimental): Once weekly
  Interventions: Drug: OSI-027
- Schedule 3 (Experimental): Once daily
  Interventions: Drug: OSI-027

INTERVENTIONS:
Drug: OSI-027 — Administered orally

SUMMARY:
The primary objective of this study is to determine the maximum tolerated dose (MTD) and to establish the recommended phase 2 dose of oral OSI-027 when administered via 3 schedules, namely, intermittent, weekly, and continuous in patients with advanced solid tumors or lymphoma, namely, intermittent, weekly, and continuous.

DETAILED DESCRIPTION:
The study will open with Schedule 1 (S1, intermittent) with initiation of Schedule 2 (S2, weekly) and Schedule 3 (S3, continuous), which may occur in parallel after observation of clinically significant related dose limiting toxicity (DLT) in the S1 schedule. Dosing will be initiated on Day 1 with intermittent weekly dosing continuing for 21 days (1 Treatment Period). Expansion of Dose Escalation Cohorts may occur for S1 and S2 at the recommended phase 2 dose level(s) and a Biomarker Expansion Cohort may be opened in S1 and/or S2.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented malignancy (solid tumor or lymphoma)
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2
* Predicted life expectancy of at least 3 months
* Adequate hematopoietic and hepatic function, and normal renal function
* Fasting glucose <7mmol/L at baseline
* Left ventricular ejection fracture (LVEF) by Multiple gated acquisition scan (MUGA)≥ 60%
* Practice effective contraceptive measures throughout study
* Verbal and written informed consent
* Prior therapy:

  * Chemotherapy, minimum of 3 weeks and recovered from any treatment-related toxicities (except for alopecia, and grade 1 neurotoxicity) prior to registration
  * Hormonal, discontinued prior to registration
  * Radiation, minimum of 21 days and recovered from toxic effects prior to registration
  * Surgery, provided wound healing has occurred

Exclusion Criteria:

* History of significant cardiac disease unless well controlled
* Discontinuation from prior therapy due to cardiac toxicity
* Active or uncontrolled infections
* Serious illness or medical condition that could interfere with study participation
* History of any psychiatric condition that might impair understanding or compliance
* Documented history of diabetes mellitus
* Pregnant or breastfeeding females
* Unstable symptomatic brain metastases, that require steroid or that have required radiation in the last 28 days
* Chronic systemic steroid use for cancer related condition
* History of allergic reactions
* Patients with cataract who are expected to undergo surgery within 6 months of registration
* Use of drugs causing QT interval prolongation within 14 days prior to dosing
* Patients with clinically significant electrolyte imbalances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 21 days

SECONDARY OUTCOMES:
Safety profile of OSI-027 | up to 5 years
Pharmacokinetic profile of OSI-027 | up to 23 days
Preliminary pharmacodynamic relationship with OSI-027 systemic exposure | up to 23 days
Preliminary antitumor activity of OSI-027 | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (3):
- Karmanos Cancer Institute, Detroit, Michigan, United States
- University Hospitals Leuven, Leuven, Belgium
- Royal Mardsen Hospital, Sutton, Surrey, United Kingdom